CLINICAL TRIAL: NCT06207565
Title: Clinical and Radiographic Evaluation of Immediate Implant Placement Utilizing Vestibular Flap Versus Single Flap Approach With Bone Graft in Anterior Maxilla: A Randomized Clinical Trial
Brief Title: Immediate Implant Placement Utilizing Vestibular Flap Versus Single Flap Approach With Bone Graft
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Responsible Party: Principal Investigator, Ahmed Abo El Futtouh, Clinical director of implant speciality program, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDCE.N6
Record Dates: First submitted 2023-12-17; First posted 2024-01-17 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Immediate Implant Placement
Keywords: Immediate implant placement; Anterior Maxilla; Vestibular flap; single flap approach

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vestibular Flap Group (Experimental): Vestibular Flap with immediate implant placement, bone graft and customized healing abutment.
  Interventions: Procedure: Vestibular Flap Group
- Single Flap Approach group (Active Comparator): Single Flap approach with immediate implant placement, bone graft and customized healing abutment.
  Interventions: Procedure: Single Flap Approach group

INTERVENTIONS:
Procedure: Vestibular Flap Group — Achieving the vestibular flap, a 1-cm long horizontal vestibular access incision using a 15c blade 3-4mm apical to the mucogingival junction of the hopeless tooth, exposing the alveolar bone. Flap dissection in a coronal direction to detach the periosteum is completed, forming a sub-periosteal tunnel.
  Arms: Vestibular Flap Group
Procedure: Single Flap Approach group — A modified envelope flap originally reported as an access flap for single implant insertion in areas of esthetic relevance will be performed. A sulcular incision on the labial aspect extending at least one tooth mesial and distal to the implant site (permitting enough accessibility for bone augmentation) is done. The flap is reflected by performing a split-thickness flap elevation starting from the interproximal incisions, leaving the anatomical papillae in situ. While the full-thickness flap elevation is performed on the labial aspect of the included surgical area, starting at the sulcus, and reaching at least 3 mm apical to the bone crest.
  Arms: Single Flap Approach group

SUMMARY:
Due to the evolution of esthetic implant dentistry and tissue regeneration (hard and soft tissue), flap design plays a crucial role in the maintenance and regeneration of the marginal soft tissue and interdental papillae around dental implants. The present study aims to compare soft and hard tissue changes following immediate implant placement with ridge augmentation using the vestibular flap versus single flap approach.

DETAILED DESCRIPTION:
Achieving and maintaining optimal esthetics around maxillary anterior single implants is a demanding task. Despite the high success rates achieved with osseointegrated implants, inevitable loss of soft and hard tissue following tooth extraction often results in compromised vertical and horizontal dimensions of the peri-implant soft tissue in terms of esthetics. Various surgical techniques have been advocated to overcome the expected alveolar ridge dimensional changes in immediate implant placement, including the use of connective tissue grafts, bone grafts, flapless implant placement protocol and the different flap designs .

Different flap designs available include vestibular incision, papilla sparing, envelope, triangular, and trapezoidal. Selection of the ideal flap design is case dependent, and is based on several factors such as, smile line, gingival biotype, width of the edentulous area, and the proposed treatment plan. It has also been reported that flapless implant placement is a predictable procedure with a high success rate and less patient discomfort, minimizing the overall procedure time, postoperative pain, and inflammation. However, flapless surgery has been regarded as a technique with limitations regarding bone augmentation.

Therefore, cases with labial bone defects during immediate implant placement require flap mobilization to achieve the needed coverage for ridge augmentation, despite of the proposed drawbacks to flap reflection, such as the increased postoperative sequelae, recovery time, and reduced blood supply after flap adaptation. A single flap approach, a modified form of the envelope flap, has been suggested as an alternative to allow for ridge augmentation in esthetic immediate implant cases with labial bone defects. Whereas the vestibular incision, one horizontal full-thickness incision in the vestibule is considered a minimally invasive aesthetic ridge augmentation technique away from the gingival margin and sulcus, intending to maintain the volume and contour of the supra crestal soft tissue.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have one non-restorable maxillary anterior (Canine to Canine region) with sound adjacent teeth.
* Intact thick biotype gingival tissue with at least 2mm band of keratinized tissue.
* Buccal bone thickness less than 1mm assessed in CBCT with good apical bone for implant primary stability.
* Good oral hygiene
* Patient accepts to provide an informed consent.

Exclusion Criteria:

* Smokers
* Pregnant and lactating females.
* Medically compromised patients.
* Patients with active infection related at the site of implant/bone graft placement.
* Patients with untreated active periodontal diseases.
* Patients with parafunctional habits.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Volumetric analysis of labial contour | 12 months
  To evaluate tissue volume changes, Intra oral scans of the esthetic zone will be obtained. Changes in the soft tissue profile will be calculated as the difference between the digitized surface outline of the different profiles at the given time of maturation of the site. All the images recorded by the intra-oral scanner will be transmitted to a 3D viewer software (Exocad Gmbh) to assess and compare the linear and volumetric changes in the labial soft tissue contour in comparison to the original, at 2, 4 and 6 mm from the pre-operative gingival margin. All the scans will be superimposed to the pre-operative scan using 3-point alignment method that ensure standardization of the images.

SECONDARY OUTCOMES:
Labio-palatal bone width | 12 months
  Two CBCT scans will be attained, primary (preoperative) scan (T0) and a secondary (Postoperative) scan 12 months after. In order to ensure standardization and reproducibility of the CBCT cross sectional images that will be used in this study, superimposition of DICOM sets of each patient using Fusion module of Ondemand 3D App software will be done (Koerich et al., 2016). This 3D superimposition technique allows for sub-voxel accuracy and highly strong registration. Both files will be loaded in the Fusion module at the same time, first manual registration will be done by approximation of the secondary scan to the primary one in axial, sagittal and coronal cuts, then automatic registration by the software. The labiopalatal width will be measured at 2 points; 2 mm apical to the crest of the palatal bone and 5mm apical to the 1st line
Mid facial recession | 12 months
  Will be measured in mm from the intraoral scans at T1, T2, T3 and compared to that of T0. The reference point will be the most apical part of the midfacial gingival level.
Interdental papillae height | 12 months
  Will be measured in mm from the intraoral scans at T1, T2, T3 and compared to that of T0. Mesial and distal papillae will be evaluated individually.

IPD SHARING:
Plan to Share IPD: No